CLINICAL TRIAL: NCT05413603
Title: Shock Wave Lithotripsy Using Fluoroscopic Versus Ultrasonic Localization for Pediatric Renal Stones.
Brief Title: Shock Wave Lithotripsy Using Fluoroscopic Versus Ultrasonic Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mahmoud Moubarak
Record Dates: First submitted 2022-05-19; First posted 2022-06-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Stone, Kidney; Child, Only
Keywords: pediatric renal stones; ultrasound shock waves; fluoroscope.
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluoroscopic focus Shock wave lithotripsy (Active Comparator): Shock wave lithotripsy, accurate localization of the shock waves is performed by the fluoroscope (FS) to fully focus the shock waves on the stone
  Interventions: Procedure: ultrasonic focus Shock wave lithotripsy; Procedure: fluoroscopic focus Shock wave lithotripsy
- ultrasonic focus Shock wave lithotripsy (Active Comparator): Shock wave lithotripsy, accurate localization of the shock waves is performed by the ultrasound (US), to fully focus the shock waves on the stone
  Interventions: Procedure: ultrasonic focus Shock wave lithotripsy; Procedure: fluoroscopic focus Shock wave lithotripsy

INTERVENTIONS:
Procedure: ultrasonic focus Shock wave lithotripsy — successful Shock wave lithotripsy , accurate localization of the shock waves is performed by ultrasound (US) to fully focus the shock waves on the stone
Procedure: fluoroscopic focus Shock wave lithotripsy — successful Shock wave lithotripsy , accurate localization of the shock waves is performed by fluoroscope (FS) to fully focus the shock waves on the stone

SUMMARY:
Epidemiological studies have shown a progressive increase in the incidence of pediatric urolithiasis over the past few decades.

DETAILED DESCRIPTION:
Pediatric stone disease is considered endemic in developing nations including Turkey, Pakistan, and eastern countries. The introduction of SWL by Chaussy et al. in the early 1980s revolutionized the management of upper urinary tract calculus disease.

Reports of successful SWL in children were first published in 1986; then several reports showed safety, and stone-free rates comparable with those of adults. For successful SWL, accurate localization of the shock waves is performed by ultrasound (US) or fluoroscope (FS) to fully focus the shock waves on the stone

ELIGIBILITY:
Inclusion Criteria:

* Children (2-16) years of age with radiopaque renal pelvic stones less than 20 mm

Exclusion Criteria:

1. Previous percutaneous nephrolithotripsy at the same side.
2. Previous renal exploration for stones at the same side.
3. Positive urinary culture.
4. Calyceal stones

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Lithotripsy or nephrolithotripsy by Shock waves | from baseline to 3 months after the Lithotripsy date.
  Incidence of success of Nephrolithotripsy by using Fluoroscopic shock waves or Ultrasonic shock waves in pediatric renal pelvic stones.

SECONDARY OUTCOMES:
Complications of shockwave lithotripsy | through study completion, an average of 1 year
  to evaluate postoperative complications of the lithotripsy as :
  1. Incidence of Hematuria
  2. Incidence of Fever
  3. Incidence of UTI
  4. Serum creatinine level in blood
  5. Rate of hydronephrosis

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Moubarak, Resident, Principal Investigator — Urology department - faculty of medicine, South Valley university.
Locations (1):
- Urology department - faculty of medicine, South Valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided